CLINICAL TRIAL: NCT01348009
Title: A Phase I-II Study of Tesetaxel Plus Capecitabine and Cisplatin in Subjects With Advanced Gastric Cancer
Brief Title: Tesetaxel Plus Capecitabine and Cisplatin in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOPK105
Record Dates: First submitted 2011-04-18; First posted 2011-05-05 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Gastric Carcinoma
Keywords: Gastric cancer; First-line therapy; Tesetaxel; Taxane; Capecitabine; Oral fluoropyrimidine; Cisplatin; Platinum
MeSH Terms: conditions — Stomach Neoplasms | interventions — tesetaxel; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tesetaxel-capecitabine-cisplatin (Experimental)
  Interventions: Drug: Tesetaxel-capecitabine-cisplatin

INTERVENTIONS:
Drug: Tesetaxel-capecitabine-cisplatin — Phase 1: Tesetaxel orally on Day 1 of each cycle at dose of 18, 21, 24, or 27 mg/m2. If no dose-limiting toxicity, at least 3 subjects will be treated at each dose level until the maximum tolerated dose or the maximum dose of 27 mg/m2 is reached. At each tesetaxel dose level, capecitabine orally at a dose of 2000 mg/m2/day (administered in 2 equally divided doses) on Day 1-Day 14 and cisplatin intravenously at a dose of 60 mg/m2 on Day 1.
  Phase 2: Tesetaxel orally on Day 1 of each cycle at dose determined in Phase 1. Capecitabine orally at a dose of 2000 mg/m2/day (administered in 2 equally divided doses) on Day 1-Day 14 and cisplatin intravenously at a dose of 60 mg/m2 on Day 1.
  Other Names: DJ-927; Xeloda; CDDP; Platinol; Platinol-AQ

SUMMARY:
Cisplatin, an intravenously administered platinum agent, in combination with an intravenously administered taxane and capecitabine has been shown to improve time to disease progression and overall survival in previously untreated patients with gastric cancer.

This study is being performed to evaluate an orally administered taxane (tesetaxel) in combination with cisplatin and capecitabine in previously untreated patients with gastric cancer.

ELIGIBILITY:
Primary Inclusion Criteria:

* At least 20 years of age
* Histologically or cytologically confirmed gastric carcinoma, including gastric or gastroesophageal-junction adenocarcinoma.
* Measurable disease (revised RECIST) based on computed tomography, or nonmeasurable disease
* Previously untreated, unresectable advanced (M0) or unresectable metastatic (M1) disease except for prior adjuvant (or neo-adjuvant) chemotherapy.
* ECOG performance status 0 or 1
* At least 4 weeks and recovery from effects of prior major surgery
* Adequate bone marrow, hepatic, and renal function

Primary Exclusion Criteria:

* Operable gastric or gastroesophageal-junction cancer
* Known brain metastasis
* Second cancer
* Previous adjuvant or neo-adjuvant chemotherapy with capecitabine and cisplatin in combination. (Previous adjuvant or neo-adjuvant monotherapy with capecitabine or S-1 or therapy with S-1 and cisplatin in combination or 5-FU and cisplatin in combination is allowed.)
* Uncontrolled diarrhea
* Nausea or vomiting for at least 3 consecutive days within the 14 days prior to registration despite the administration of standard antiemetic therapy
* Symptomatic peripheral neuropathy ≥ Grade 2
* Malabsorption syndrome or other disease that significantly affects gastrointestinal function
* Other uncontrolled systemic illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate (in Phase 2 portion of study) | 6 months from the date of first dose of study medication

SECONDARY OUTCOMES:
Recommended dose of tesetaxel for Phase 2 (in Phase 1 portion of study) | Up to 21 days after first dose of study medication
  The dose of tesetaxel in mg/m2 will be determined for Phase 2 based on the occurrence of dose-limiting toxicities in Phase 1.
Response rate, as defined in revised RECIST (in Phase 2 portion of study) | Up to 12 months following the date of first dose of study medication
Duration of response (in Phase 2 portion of study) | Up to 12 months following the date of first dose of study medication
Rate of responses at least 3 months in duration (in Phase 2 portion of study) | Up to 12 months following the date of first dose of study medication
Disease control rate, which is defined as the percentage of patients with a response of any duration or stable disease at least 6 weeks in duration (in Phase 2 portion of study) | Up to 12 months following the date of first dose of study medication
Durable response rate, which is defined as the percentage of patients with a response at least 6 months in duration (in Phase 2 portion of study) | Up to 12 months following the date of first dose of study medication
Progression-free survival (in Phase 2 portion of study) | Up to 12 months following the date of first dose of study medication
Overall survival (in Phase 2 portion of study) | Up to 12 months following the date of first dose of study medication
Percentage of patients with adverse events (in Phase 1 and Phase 2 portions) | Up to 30 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Rha, MD, PhD, Principal Investigator — Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Yonsei Cancer Center, Yonsei University College of Medicine, Seoul, South Korea